CLINICAL TRIAL: NCT01379235
Title: Association Between Pilatis Exercise, Balance and Stability Measurements, and Quality of Life Among Elderly Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MMC105809KCTIL
Record Dates: First submitted 2011-02-15; First posted 2011-06-23 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2012-06

CONDITIONS: Quality of Life; Accidental Falls
Keywords: independent 65 years old and above

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental): Intervention group: will receive 12 weeks of pilatis exercise 3 times a week.
  Interventions: Other: Pilatis exercise
- control group (Other): The control group will be offered the same intervention (pilatis exercise) at the end of the study period.
  Interventions: Other: Pilatis exercise

INTERVENTIONS:
Other: Pilatis exercise — 12 weeks of pilatis exercise 3 times a week.

SUMMARY:
Background: The elderly population in western countries and in Israel is constantly growing. Falls are one of the common problems among this population. Thus there is a need for falls prevention exercise program to be offered in the different settings elderly reside. Most methods for physical exercise are dedicated to muscle strengthening and improving balance by strengthening external muscles. Pilatis exercise program focuses mainly on strengthening the in-depth muscles. The advantage of this method is in its simplicity and availability. This method is suitable also for special populations as patients in acute hospitalization. In this study, the investigators will evaluate if the pilatis exercise can improve balance of elderly population. Physical exercise usually improves the mood. Like any physical exercise, Pilatis exercise has a mental advantage, therefore, this study will also examine if pilatis exercise can improve quality of life of elderly population.

Working hypothesis and aims: Pilatis exercise will improve balance and stability measurements, and quality of life among elderly population.

Methods: Randomized, prospective study among elderly patients aged 65 and above belonging to Clalit Health Services primary care clinic . Participants of the intervention and control group will receive a brochure that will include nutrition and healthy life style recommendations. Intervention group: will receive 12 weeks of pilatis exercise 3 times a week. The control group will be offered the same intervention at the end of the study period. Balance evaluation will be performed using the: Tinetti Balance Gait Scale, Berg Balance Scale, Multidirectional Reach Test, Timed Up and Go, Step execution test. The SF-36 questionnaire will be use to evaluate quality of life.

Importance: This study will examine the influence of pilatis exercise on balance among the elderly. If findings will determine that pilatis does improve balance in the elderly, the investigators can further examine pilatis's influence on falls prevention, and minimizing falls damages.

Probable implications to the welfare and health of the aged population:

Improving balance, falls preventing and minimizing falls damages among elderly; improvement in elderly quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Man and Women aged 65 years old and above
* Able to walk independently without devices (cane is exceptable)

Exclusion Criteria:

1. Unstable diseases (unstable angina; heart failure- NIHA 3 or 4; lung disease with shortness of breath on light effort; end stage liver and kidney diseases; terminal malignant diseases)
2. MMSE less then 24
3. After hip or knee surgery
4. After lower limb amputation
5. Neurological diseases with significant gait and balance instability.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 88 (Actual)
Dates: Start 2012-01; Primary Completion 2012-10 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
postural stability test | 3 months
  Statistically significance difference in postural stability test will be found when comparing pre and post intervention results in the intervention group of the Step execution test. This outcome is a combination of the variables: elliptical area(mm2), sway velocity (mm/s), mediolateral sway (mm)and anterior posterior sway (mm).

CONTACTS AND LOCATIONS:
Overall Officials: Yan Press, MD, Principal Investigator — Ben-Gurion University of the Negev
Locations (1):
- Clalit Health Services (HMO), Beersheba, Israel